CLINICAL TRIAL: NCT03328585
Title: Telemedicine vs. In-person Delivery of Cognitive Behavioral Treatment of Insomnia: a Mixed Methods Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 827001
Record Dates: First submitted 2017-10-20; First posted 2017-11-01 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Insomnia Disorder
Keywords: CBT-I; Telemedicine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT-I in person (Active Comparator)
  Interventions: Behavioral: CBT-I in person
- CBT-I via telemedicine (Experimental)
  Interventions: Behavioral: CBT-I via Telemedicine
- Waitlist Control (Other): Patients in this arm will receive in person CBT-I treatment after conclusion of the study.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: CBT-I in person — 6 weeks of CBT-I in person, one 1-hour long session per week
  Arms: CBT-I in person
Behavioral: CBT-I via Telemedicine — 6 weeks of CBT-I via telemedicine, one 1-hour long session per week
  Arms: CBT-I via telemedicine
Other: No intervention — Patients in this arm will receive no intervention but will receive CBT-I treatment after conclusion of the study
  Arms: Waitlist Control

SUMMARY:
Cognitive behavioral therapy for insomnia (CBT-I) has been the 'gold standard' for the treatment of insomnia. There is a need to increase access to treatment, particularly for patients in more rural locations where providers may be scarce. One solution is to utilize telemedicine which is "the use of electronic communications to provide and support health care when distance separates the provider from the patient." So the purpose of the study is to determine if receiving CBT-I by video teleconferencing works just as well as in-person treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet current DSM5 criteria for Insomnia Disorder as determined by clinician interview
* ISI score greater than 14, with self-reported duration of insomnia of at least 3 months
* Ability to read and speak English
* Own a personal computer with an internet connection sufficient to utilize the SleepTM and REDCap platform
* BMI less than 30
* Between the ages of 21-50

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Individuals with an untreated sleep disorder other than insomnia (Individuals with sleep apnea who are adherent with CPAP treatment (average 4 hours use per night) will be eligible to participate)
* A clinically unstable medical condition as defined by a new diagnosis or change in medical management in the previous 2 months
* Individuals with substance abuse/dependence, bipolar disorder, delirium, dementia, amnestic disorder, schizophrenia, and other psychotic disorders
* Individuals with prominent current suicidal or homicidal ideation
* Unable to perform tests due to inability to communicate verbally, inability to read and write; less than a 5th grade reading level; visual, hearing, or cognitive impairment
* Any use of medications or OTC products that might impact sleep or metabolism

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in ISI scores | Once at baseline assessment and once again at follow-up after CBT-I intervention approximately 9 weeks later
  Total score on the Insomnia Severity Index (0-28)

SECONDARY OUTCOMES:
Change in actigraphic sleep efficiency | Patients will wear the wristband for a week during sleep baseline assessment and again for a week at follow-up, approximately 8 weeks later
  Measured using an actigraph wristband

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gehrman P, Gunter P, Findley J, Frasso R, Weljie AM, Kuna ST, Kayser MS. Randomized Noninferiority Trial of Telehealth Delivery of Cognitive Behavioral Treatment of Insomnia Compared to In-Person Care. J Clin Psychiatry. 2021 Aug 24;82(5):20m13723. doi: 10.4088/JCP.20m13723. PMID 34428360